CLINICAL TRIAL: NCT03500393
Title: A Remotely Supervised Exercise Program for Lung Cancer Patients Undergoing Chemoradiation
Brief Title: A Remotely Supervised Exercise Program for Lung Cancer Patients Undergoing Chemoradiation (REM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasibility of study recruitment
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Kathleen Lyons, Scientist, Psychiatry Research, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D18012
Record Dates: First submitted 2018-03-16; First posted 2018-04-18 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the remotely supervised exercise (REM) or the unsupervised exercise (UNSUP) arm upon completion of the baseline assessment battery.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blind to study hypotheses, data collector will be blind to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unsupervised Exercise (UNSUP) (Active Comparator): The control condition represents a minimalist intervention that could occur in any setting: (1) enthusiastic provision on an exercise prescription and (2) provision of a fitness device (i.e., the Garmin VivioActive) that can help participants track their exercise engagement. Participants are instructed in how to use the device to track their adherence to the exercise prescription.
  Interventions: Behavioral: Unsupervised Exercise (UNSUP)
- Remotely Supervised Exercise (REM) (Experimental): The REM program is designed to function as an Acceptance-based health coaching intervention and will utilize theory-based behavior change techniques (i.e., goal setting/action planning, self-monitoring, receiving feedback, and reviewing relevant goals in the light of feedback) to promote adoption and adherence to the exercise prescription.
  Interventions: Behavioral: Remotely Supervised Exercise (REM)

INTERVENTIONS:
Behavioral: Remotely Supervised Exercise (REM) — REM is designed to follow in the tradition of stepped care behavioral interventions. As such, participants who are successfully engaging in the prescribed exercise are provided minimal and automated encouragement and praise. Participants who demonstrate less adherence are given interventions that are tailored in content and intensity, depending on the level of success and the nature of the barriers to success
  Arms: Remotely Supervised Exercise (REM)
Behavioral: Unsupervised Exercise (UNSUP) — The control condition represents a minimalist intervention that could occur in any setting: (1) enthusiastic provision on an exercise prescription and (2) provision of a fitness device (i.e., the Garmin VivioActive) that can help participants track their exercise engagement. Participants are instructed in how to use the device to track their adherence to the exercise prescription.
  Arms: Unsupervised Exercise (UNSUP)

SUMMARY:
The purpose of this study is to conduct a pilot randomized controlled trial (RCT) evaluating the feasibility and potential effectiveness of a remotely supervised exercise program (REM) in promoting adherence to an exercise prescription before and during chemoradiation.

DETAILED DESCRIPTION:
The research team adopts an overtly pragmatic approach where our design choices are made to enhance external validity and create a parsimonious intervention that can be integrated into busy clinical practices. This is a pilot study and is not designed to definitively provide evidence for a treatment effect, but rather to establish feasibility and to optimize the intervention and study procedures in preparation for a larger trial. We will conduct a pilot RCT comparing a remotely supervised exercise program (REM) to an unsupervised exercise program (UNSUP). Data will be collected upon enrollment (T0; at least 2 weeks prior to beginning chemoradiation), immediately prior to chemoradiation (T1), immediately post-chemoradiation (T2) and 1-month post-chemoradiation (T3).

ELIGIBILITY:
Inclusion Criteria:

* Are over the age of 18 and diagnosed with Stage IIa to IIIb lung cancer;
* Definitive treatment with chemoradiation with weekly carboplatin and paclitaxel concurrent with radiation is planned to begin in no less than 2 weeks;
* Have an Apple or Android device with capacity to install a fitness device app and access to either WiFi or cellular service;
* Are English-speaking and able to provide voluntary, written consent;
* Able to tolerate chemoradiation as indicated by Zubrod/ECOG Performance Status 0-1; CBC/differential obtained within 14 days prior to registration on study, with adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl;Adequate renal function within 14 days prior to registration, defined as creatinine clearance must be at least 35 ml/min; Adequate hepatic function within 14 days prior to registration, defined as total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution and ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution; No prior thoracic radiation therapy;

Exclusion Criteria:

* Life expectancy of < 12 months or are receiving hospice services;
* Psychiatric diagnosis that would require significant study modification to meet their needs such as uncontrolled severe mental illness, substance abuse, or active suicidal ideation;
* Exhibit American College of Sports Medicine contraindications to exercise which include a resting heart rate of >120bpm, blood pressure >180/100mmHg or unstable angina 40 or musculoskeletal issue preventing exercise;
* Are unable to walk 100 meters. According to our current standard of care, those participants will be referred to physical therapy for evaluation and treatment and will be excluded from the study as unsupervised exercise would not be safe;
* Less than 2 weeks to the beginning of chemoradiation;
* Physician discretion;
* Are unable to walk or to complete the 6-minute walk test. According to our current standard of care, those participants will be referred to physical therapy for evaluation and treatment and will be excluded from the study as unsupervised exercise would not be safe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention statistics | Time 3, One month after completing chemoradiation
  Number of participants enrolled/number of patients eligible; Number completing all data collection/Number enrolled; Number adhering to randomization/number enrolled; Number withdrawn/number enrolled

SECONDARY OUTCOMES:
Minutes spent in exercise | Time 3, One month after completing chemoradiation
  Objective measure of adherence to exercise prescription; collected from fitness device
6-minute walk test | Time 3, One month after completing chemoradiation
  Observational measure of aerobic capacity (measures how far you can walk in six minutes)
Timed up-and-go test | Time 3, One month after completing chemoradiation
  Observational measure of functional capacity/balance and agility (measures how long it takes to rise walk three meters, turn and sit)
Five times sit-to-stand test | Time 3, One month after completing chemoradiation
  Observational measure of functional capacity/lower extremity strength (measures how long it take to rise from and sit down in chair five times)
Forced expiratory volume in 1 second | Time 3, One month after completing chemoradiation
  Pulmonary function will be measured by forced expiratory volume in 1 second (FEV1). This will be measured by a pulmonary medicine technician as part of the pre-chemoradiation (T0) exam and 1-month post-treatment (T3).
Diffusion capacity | Time 3, One month after completing chemoradiation
  Pulmonary function will be measured by the diffusing capacity of lungs for carbon monoxide (DLCO). This will be measured by a pulmonary medicine technician as part of the pre-chemoradiation (T0) exam and 1-month post-treatment (T3).
Forced vital capacity | Time 3, One month after completing chemoradiation
  Pulmonary function will be measured by forced vital capacity (FVC). This will be measured by a pulmonary medicine technician as part of the pre-chemoradiation (T0) exam and 1-month post-treatment (T3).
Physical Function Scale of the Patient Reported Outcomes Measurement information System (PROMIS) | Time 3, One month after completing chemoradiation
  The 10-item physical function scale of the PROMIS Item Bank36 will be administered to the participant by the research assistant. The items ask respondents to determine the degree to which health interferes with mobility and daily living tasks. The scale has an internal reliability coefficient of 0.81 and was found to correlate positively with quality of life and negatively with pain impact. Higher scores indicate better physical function.
Pittsburgh Sleep Quality Index | Time 3, One month after completing chemoradiation
  From the actigraphy data from the Garmin fitness device, we can calculate sleep onset latency (SOL), total sleep time (TST), wake after sleep onset (WASO), and sleep efficiency (SE). It is expected that increased exercise in cancer patients will follow by decreased SOL and WASO, increased TST and SE, and improvements in subjective sleep quality. The Pittsburgh Sleep Quality Index (PSQI) is a widely used measure of sleep quality, in the time frame of 2 weeks prior to the assessment. PSQI assesses a range of sleep disturbances, including symptoms of insomnia, symptoms of sleep-related breathing disorders, use of sleep medications, etc. PSQI score over 5 is indicative of significant sleep disturbances. We would expect that PSQI score would decrease following increased exercise in cancer patients.
Functional Assessment of Cancer Therapy-fatigue scale | Time 3, One month after completing chemoradiation
  The Functional Assessment of Cancer Treatment- Fatigue (FACT-F) instrument will be used to measure quality of life and, specifically, effects of cancer-related fatigue upon quality of life .37 The FACT-F is a 40-item self-report measure of health-related quality of life specifically designed for cancer patients. The first 27 items of the tool represent the general version of the FACT (FACT-G) which assesses perceived well-being in physical, social, emotional, and functional domains. The remainder of the tool addresses concerns directly relevant to fatigue. Higher scores indicate higher quality of life.
Dose reductions | Time 3, One month after completing chemoradiation
  Medical record audits will be conducted to determine the degree to which participants received the prescribed regimen of chemoradiation (performed at T2).
Grip strength | Time 3, one month after completing chemoradiation
  Grip strength has been found to effectively identify people with clinically significant weakness that correlates with disability.60 Using a JAMAR Handheld Dynamometer, the subject will hold the device in their dominant hand, with the arm at right angles and the elbow by the side of the body. No other body movement is allowed. The subject squeezes the dynamometer with maximum isometric effort and maintained for about 5 seconds. The subject should be strongly encouraged to give maximum effort. The best result from several trials for each hand is recorded with at least 15 seconds recovery between each effort.

OTHER OUTCOMES:
Physical Activity Acceptance Questionnaire | Time 2, Assessment immediately after completing chemoradiation
  To explore the hypothesized mechanism underlying the effect of the intervention on exercise adherence we will measure psychological flexibility. The Physical Activity Acceptance Questionnaire (PAAQ)61 is a 10-item scale used to measure a person's ability to accept physical and psychological discomfort in the context of exercise. All items on the PAAQ are rated on a 7-point Likert scale scored, 1 = strongly disagree to 7 = strongly agree. Psychological flexibility is a stance of openness to the present experience (i.e., one's thoughts and feelings) without attempts to modify, suppress, or terminate that experience in any way. Responses to these items were summed to yield PAAQ total scores (at each time point) ranging from 10 - 70 where higher scores represent stronger experiential acceptance.
Lymphocyte subsets | Time 3, One month after completing chemoradiation
  To explore the possible mechanisms underlying the effect of exercise, we will collect peripheral blood samples to analyze lymphocyte subsets, cytokines, and stress hormones. Flow cytometry will be used to analyze Total CD3+cells, Total CD4+ and CD8 cells and Treg populations in peripheral blood. Plasma/Serum will be stored for batch multi-plex ELISA for pro-and anti-inflammatory cytokine and stress hormone analyses
Inflammatory cytokines | Time 3, One month after completing chemoradiation
  To explore the possible mechanisms underlying the effect of exercise, we will collect peripheral blood samples to analyze lymphocyte subsets, cytokines, and stress hormones. Flow cytometry will be used to analyze Total CD3+cells, Total CD4+ and CD8 cells and Treg populations in peripheral blood. Plasma/Serum will be stored for batch multi-plex ELISA for pro-and anti-inflammatory cytokine and stress hormone analyses
Stress hormones | Time 3, One month after completing chemoradiation
  To explore the possible mechanisms underlying the effect of exercise, we will collect peripheral blood samples to analyze lymphocyte subsets, cytokines, and stress hormones. Flow cytometry will be used to analyze Total CD3+cells, Total CD4+ and CD8 cells and Treg populations in peripheral blood. Plasma/Serum will be stored for batch multi-plex ELISA for pro-and anti-inflammatory cytokine and stress hormone analyses

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Lyons, ScD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Cancer Society. Cancer Facts and Figures 2016. Atlanta, GA2016
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Margaritora S, Cesario A, Cusumano G, Cafarotti S, Corbo GM, Ferri L, Ceppi M, Meacci E, Valente S, D'Angelillo RM, Russo P, Porziella V, Bonassi S, Pasqua F, Sterzi S, Granone P. Is pulmonary function damaged by neoadjuvant lung cancer therapy? A comprehensive serial time-trend analysis of pulmonary function after induction radiochemotherapy plus surgery. J Thorac Cardiovasc Surg. 2010 Jun;139(6):1457-63. doi: 10.1016/j.jtcvs.2009.10.023. Epub 2010 Apr 2. PMID 20363001
- [Background] Pasqua F, Biscione G, Crigna G, Auciello L, Cazzola M. Combining triple therapy and pulmonary rehabilitation in patients with advanced COPD: a pilot study. Respir Med. 2010 Mar;104(3):412-7. doi: 10.1016/j.rmed.2009.10.005. Epub 2009 Nov 4. PMID 19892540
- [Background] Cesario A, Ferri L, Galetta D, Pasqua F, Bonassi S, Clini E, Biscione G, Cardaci V, di Toro S, Zarzana A, Margaritora S, Piraino A, Russo P, Sterzi S, Granone P. Post-operative respiratory rehabilitation after lung resection for non-small cell lung cancer. Lung Cancer. 2007 Aug;57(2):175-80. doi: 10.1016/j.lungcan.2007.02.017. Epub 2007 Apr 17. PMID 17442449
- [Background] Jackson W, Alexander N, Schipper M, Fig L, Feng F, Jolly S. Characterization of changes in total body composition for patients with head and neck cancer undergoing chemoradiotherapy using dual-energy x-ray absorptiometry. Head Neck. 2014 Sep;36(9):1356-62. doi: 10.1002/hed.23461. Epub 2013 Nov 21. PMID 23970480
- [Background] Carli F, Scheede-Bergdahl C. Prehabilitation to enhance perioperative care. Anesthesiol Clin. 2015 Mar;33(1):17-33. doi: 10.1016/j.anclin.2014.11.002. Epub 2015 Jan 9. PMID 25701926
- [Background] Silver JK, Baima J. Cancer prehabilitation: an opportunity to decrease treatment-related morbidity, increase cancer treatment options, and improve physical and psychological health outcomes. Am J Phys Med Rehabil. 2013 Aug;92(8):715-27. doi: 10.1097/PHM.0b013e31829b4afe. PMID 23756434
- [Background] Carli F, Zavorsky GS. Optimizing functional exercise capacity in the elderly surgical population. Curr Opin Clin Nutr Metab Care. 2005 Jan;8(1):23-32. doi: 10.1097/00075197-200501000-00005. PMID 15585997
- [Background] Jones LW, Watson D, Herndon JE 2nd, Eves ND, Haithcock BE, Loewen G, Kohman L. Peak oxygen consumption and long-term all-cause mortality in nonsmall cell lung cancer. Cancer. 2010 Oct 15;116(20):4825-32. doi: 10.1002/cncr.25396. PMID 20597134
- [Background] Tarumi S, Yokomise H, Gotoh M, Kasai Y, Matsuura N, Chang SS, Go T. Pulmonary rehabilitation during induction chemoradiotherapy for lung cancer improves pulmonary function. J Thorac Cardiovasc Surg. 2015 Feb;149(2):569-73. doi: 10.1016/j.jtcvs.2014.09.123. Epub 2014 Oct 5. PMID 25451483
- [Background] Yeh SH, Lai HL, Hsiao CY, Lin LW, Chuang YK, Yang YY, Yang KD. Moderate physical activity of music aerobic exercise increases lymphocyte counts, specific subsets, and differentiation. J Phys Act Health. 2014 Sep;11(7):1386-92. doi: 10.1123/jpah.2012-0508. Epub 2013 Dec 20. PMID 24368695
- [Background] Wang R, Liu J, Chen P, Yu D. Regular tai chi exercise decreases the percentage of type 2 cytokine-producing cells in postsurgical non-small cell lung cancer survivors. Cancer Nurs. 2013 Jul-Aug;36(4):E27-34. doi: 10.1097/NCC.0b013e318268f7d5. PMID 23051870
- [Background] Silver JK. Cancer prehabilitation and its role in improving health outcomes and reducing health care costs. Semin Oncol Nurs. 2015 Feb;31(1):13-30. doi: 10.1016/j.soncn.2014.11.003. Epub 2014 Dec 3. PMID 25636392
- [Background] Kleinman MS, Mold JW. Defining the components of the research pipeline. Clin Transl Sci. 2009 Aug;2(4):312-4. doi: 10.1111/j.1752-8062.2009.00119.x. PMID 20443910
- [Background] Holmes MD, Chen WY, Feskanich D, Kroenke CH, Colditz GA. Physical activity and survival after breast cancer diagnosis. JAMA. 2005 May 25;293(20):2479-86. doi: 10.1001/jama.293.20.2479. PMID 15914748
- [Background] Jones LW, Viglianti BL, Tashjian JA, Kothadia SM, Keir ST, Freedland SJ, Potter MQ, Moon EJ, Schroeder T, Herndon JE 2nd, Dewhirst MW. Effect of aerobic exercise on tumor physiology in an animal model of human breast cancer. J Appl Physiol (1985). 2010 Feb;108(2):343-8. doi: 10.1152/japplphysiol.00424.2009. Epub 2009 Dec 3. PMID 19959769
- [Background] Moore SC, Lee IM, Weiderpass E, Campbell PT, Sampson JN, Kitahara CM, Keadle SK, Arem H, Berrington de Gonzalez A, Hartge P, Adami HO, Blair CK, Borch KB, Boyd E, Check DP, Fournier A, Freedman ND, Gunter M, Johannson M, Khaw KT, Linet MS, Orsini N, Park Y, Riboli E, Robien K, Schairer C, Sesso H, Spriggs M, Van Dusen R, Wolk A, Matthews CE, Patel AV. Association of Leisure-Time Physical Activity With Risk of 26 Types of Cancer in 1.44 Million Adults. JAMA Intern Med. 2016 Jun 1;176(6):816-25. doi: 10.1001/jamainternmed.2016.1548. PMID 27183032
- [Background] Santa Mina D, Scheede-Bergdahl C, Gillis C, Carli F. Optimization of surgical outcomes with prehabilitation. Appl Physiol Nutr Metab. 2015 Sep;40(9):966-9. doi: 10.1139/apnm-2015-0084. Epub 2015 May 13. PMID 26300015
- [Background] Armstrong KW, Bravo-Iniguez CE, Jacobson FL, Jaklitsch MT. Recent trends in surgical research of cancer treatment in the elderly, with a primary focus on lung cancer: Presentation at the 2015 annual meeting of SIOG. J Geriatr Oncol. 2016 Sep;7(5):368-74. doi: 10.1016/j.jgo.2016.07.004. Epub 2016 Jul 25. PMID 27460994
- [Background] Singh F, Newton RU, Galvao DA, Spry N, Baker MK. A systematic review of pre-surgical exercise intervention studies with cancer patients. Surg Oncol. 2013 Jun;22(2):92-104. doi: 10.1016/j.suronc.2013.01.004. Epub 2013 Feb 19. PMID 23434347
- [Background] Sebio Garcia R, Yanez Brage MI, Gimenez Moolhuyzen E, Granger CL, Denehy L. Functional and postoperative outcomes after preoperative exercise training in patients with lung cancer: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Sep;23(3):486-97. doi: 10.1093/icvts/ivw152. Epub 2016 May 25. PMID 27226400
- [Background] Crandall K, Maguire R, Campbell A, Kearney N. Exercise intervention for patients surgically treated for Non-Small Cell Lung Cancer (NSCLC): a systematic review. Surg Oncol. 2014 Mar;23(1):17-30. doi: 10.1016/j.suronc.2014.01.001. Epub 2014 Jan 24. PMID 24529937
- [Background] Pouwels S, Fiddelaers J, Teijink JA, Woorst JF, Siebenga J, Smeenk FW. Preoperative exercise therapy in lung surgery patients: A systematic review. Respir Med. 2015 Dec;109(12):1495-504. doi: 10.1016/j.rmed.2015.08.009. Epub 2015 Aug 15. PMID 26303337
- [Background] Jones LW, Peddle CJ, Eves ND, Haykowsky MJ, Courneya KS, Mackey JR, Joy AA, Kumar V, Winton TW, Reiman T. Effects of presurgical exercise training on cardiorespiratory fitness among patients undergoing thoracic surgery for malignant lung lesions. Cancer. 2007 Aug 1;110(3):590-8. doi: 10.1002/cncr.22830. PMID 17582629
- [Background] Jones LW, Eves ND, Peterson BL, Garst J, Crawford J, West MJ, Mabe S, Harpole D, Kraus WE, Douglas PS. Safety and feasibility of aerobic training on cardiopulmonary function and quality of life in postsurgical nonsmall cell lung cancer patients: a pilot study. Cancer. 2008 Dec 15;113(12):3430-9. doi: 10.1002/cncr.23967. PMID 18988290
- [Background] Stout NL, Baima J, Swisher AK, Winters-Stone KM, Welsh J. A Systematic Review of Exercise Systematic Reviews in the Cancer Literature (2005-2017). PM R. 2017 Sep;9(9S2):S347-S384. doi: 10.1016/j.pmrj.2017.07.074. PMID 28942909
- [Background] Stene GB, Helbostad JL, Balstad TR, Riphagen II, Kaasa S, Oldervoll LM. Effect of physical exercise on muscle mass and strength in cancer patients during treatment--a systematic review. Crit Rev Oncol Hematol. 2013 Dec;88(3):573-93. doi: 10.1016/j.critrevonc.2013.07.001. Epub 2013 Aug 9. PMID 23932804
- [Background] Hoffman AJ, Brintnall RA, von Eye A, Jones LW, Alderink G, Patzelt LH, Brown JK. Home-based exercise: promising rehabilitation for symptom relief, improved functional status and quality of life for post-surgical lung cancer patients. J Thorac Dis. 2014 Jun;6(6):632-40. doi: 10.3978/j.issn.2072-1439.2014.06.08. PMID 24976984
- [Background] Weinhold M, Shimabukuro-Vornhagen A, Franke A, Theurich S, Wahl P, Hallek M, Schmidt A, Schinkothe T, Mester J, von Bergwelt-Baildon M, Bloch W. Physical exercise modulates the homeostasis of human regulatory T cells. J Allergy Clin Immunol. 2016 May;137(5):1607-1610.e8. doi: 10.1016/j.jaci.2015.10.035. Epub 2016 Jan 7. No abstract available. PMID 26774657
- [Background] Niemela M, Kangastupa P, Niemela O, Bloigu R, Juvonen T. Acute Changes in Inflammatory Biomarker Levels in Recreational Runners Participating in a Marathon or Half-Marathon. Sports Med Open. 2016 Dec;2(1):21. doi: 10.1186/s40798-016-0045-0. Epub 2016 Mar 2. PMID 27747777
- [Background] Treanor C, Kyaw T, Donnelly M. An international review and meta-analysis of prehabilitation compared to usual care for cancer patients. J Cancer Surviv. 2018 Feb;12(1):64-73. doi: 10.1007/s11764-017-0645-9. Epub 2017 Sep 12. PMID 28900822
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Mesquita R, Wilke S, Smid DE, Janssen DJ, Franssen FM, Probst VS, Wouters EF, Muris JW, Pitta F, Spruit MA. Measurement properties of the Timed Up & Go test in patients with COPD. Chron Respir Dis. 2016 Nov;13(4):344-352. doi: 10.1177/1479972316647178. Epub 2016 Jul 8. PMID 27165963
- [Background] Jones SE, Kon SS, Canavan JL, Patel MS, Clark AL, Nolan CM, Polkey MI, Man WD. The five-repetition sit-to-stand test as a functional outcome measure in COPD. Thorax. 2013 Nov;68(11):1015-20. doi: 10.1136/thoraxjnl-2013-203576. Epub 2013 Jun 19. PMID 23783372
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Sox HC, Lewis RJ. Pragmatic Trials: Practical Answers to "Real World" Questions. JAMA. 2016 Sep 20;316(11):1205-1206. doi: 10.1001/jama.2016.11409. No abstract available. PMID 27654606
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] McDermott MM, Guralnik JM, Criqui MH, Ferrucci L, Liu K, Spring B, Tian L, Domanchuk K, Kibbe M, Zhao L, Lloyd Jones D, Liao Y, Gao Y, Rejeski WJ. Unsupervised exercise and mobility loss in peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2015 May 20;4(5):e001659. doi: 10.1161/JAHA.114.001659. PMID 25994445
- [Background] Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health Psychol. 2009 Nov;28(6):690-701. doi: 10.1037/a0016136. PMID 19916637
- [Background] Carver CS, Scheier MF. Control theory: a useful conceptual framework for personality-social, clinical, and health psychology. Psychol Bull. 1982 Jul;92(1):111-35. No abstract available. PMID 7134324
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] Coughlin SS, Stewart J. Use of Consumer Wearable Devices to Promote Physical Activity: A Review of Health Intervention Studies. J Environ Health Sci. 2016 Nov;2(6):10.15436/2378-6841.16.1123. doi: 10.15436/2378-6841.16.1123. Epub 2016 Nov 30. PMID 28428979
- [Background] de Vries HJ, Kooiman TJ, van Ittersum MW, van Brussel M, de Groot M. Do activity monitors increase physical activity in adults with overweight or obesity? A systematic review and meta-analysis. Obesity (Silver Spring). 2016 Oct;24(10):2078-91. doi: 10.1002/oby.21619. PMID 27670401
- [Background] Dobkin BH, Dorsch A. The promise of mHealth: daily activity monitoring and outcome assessments by wearable sensors. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):788-98. doi: 10.1177/1545968311425908. PMID 21989632
- [Background] Mendoza L, Horta P, Espinoza J, Aguilera M, Balmaceda N, Castro A, Ruiz M, Diaz O, Hopkinson NS. Pedometers to enhance physical activity in COPD: a randomised controlled trial. Eur Respir J. 2015 Feb;45(2):347-54. doi: 10.1183/09031936.00084514. Epub 2014 Sep 26. PMID 25261324
- [Background] Kwan BM, Bryan A. In-task and post-task affective response to exercise: translating exercise intentions into behaviour. Br J Health Psychol. 2010 Feb;15(Pt 1):115-31. doi: 10.1348/135910709X433267. Epub 2009 Apr 25. PMID 19397847
- [Background] Schneider M, Dunn A, Cooper D. Affect, exercise, and physical activity among healthy adolescents. J Sport Exerc Psychol. 2009 Dec;31(6):706-23. doi: 10.1123/jsep.31.6.706. PMID 20384008
- [Background] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Goodwin CL, Forman EM, Herbert JD, Butryn ML, Ledley GS. A pilot study examining the initial effectiveness of a brief acceptance-based behavior therapy for modifying diet and physical activity among cardiac patients. Behav Modif. 2012 Mar;36(2):199-217. doi: 10.1177/0145445511427770. Epub 2011 Nov 30. PMID 22133992
- [Background] Hawkes AL, Chambers SK, Pakenham KI, Patrao TA, Baade PD, Lynch BM, Aitken JF, Meng X, Courneya KS. Effects of a telephone-delivered multiple health behavior change intervention (CanChange) on health and behavioral outcomes in survivors of colorectal cancer: a randomized controlled trial. J Clin Oncol. 2013 Jun 20;31(18):2313-21. doi: 10.1200/JCO.2012.45.5873. Epub 2013 May 20. PMID 23690410
- [Background] Stevens CJ. Get ACTive! A randomized controlled trial of feasibility and effectiveness of an acceptance-based behavioral intervention to promote exercise adoption and maintenance. 2016.
- [Background] Bower P, Gilbody S. Stepped care in psychological therapies: access, effectiveness and efficiency. Narrative literature review. Br J Psychiatry. 2005 Jan;186:11-7. doi: 10.1192/bjp.186.1.11. PMID 15630118
- [Background] Gabrielson DK, Scaffidi D, Leung E, Stoyanoff L, Robinson J, Nisenbaum R, Brezden-Masley C, Darling PB. Use of an abridged scored Patient-Generated Subjective Global Assessment (abPG-SGA) as a nutritional screening tool for cancer patients in an outpatient setting. Nutr Cancer. 2013;65(2):234-9. doi: 10.1080/01635581.2013.755554. PMID 23441610
- [Background] Vigano AL, di Tomasso J, Kilgour RD, Trutschnigg B, Lucar E, Morais JA, Borod M. The abridged patient-generated subjective global assessment is a useful tool for early detection and characterization of cancer cachexia. J Acad Nutr Diet. 2014 Jul;114(7):1088-1098. doi: 10.1016/j.jand.2013.09.027. Epub 2014 Jan 24. PMID 24462323
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Alley DE, Shardell MD, Peters KW, McLean RR, Dam TT, Kenny AM, Fragala MS, Harris TB, Kiel DP, Guralnik JM, Ferrucci L, Kritchevsky SB, Studenski SA, Vassileva MT, Cawthon PM. Grip strength cutpoints for the identification of clinically relevant weakness. J Gerontol A Biol Sci Med Sci. 2014 May;69(5):559-66. doi: 10.1093/gerona/glu011. PMID 24737558
- [Background] Butryn ML, Arigo D, Raggio GA, Kaufman AI, Kerrigan SG, Forman EM. Measuring the Ability to Tolerate Activity-Related Discomfort: Initial Validation of the Physical Activity Acceptance Questionnaire (PAAQ). J Phys Act Health. 2015 May;12(5):717-6. doi: 10.1123/jpah.2013-0338. Epub 2014 Aug 7. PMID 25106049
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005;4(4):287-291.
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Hegel MT, Lyons KD, Hull JG, Kaufman P, Urquhart L, Li Z, Ahles TA. Feasibility study of a randomized controlled trial of a telephone-delivered problem-solving-occupational therapy intervention to reduce participation restrictions in rural breast cancer survivors undergoing chemotherapy. Psychooncology. 2011 Oct;20(10):1092-101. doi: 10.1002/pon.1830. Epub 2010 Sep 5. PMID 20821373
- [Background] Lyons KD, Newman RM, Kaufman PA, Bruce ML, Stearns DM, Lansigan F, Chamberlin M, Bartels SJ, Whipple J, Hegel MT. Goal Attainment and Goal Adjustment of Older Adults During Person-Directed Cancer Rehabilitation. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205110p1-7202205110p8. doi: 10.5014/ajot.2018.023648. PMID 29426388
- [Background] Lyons KD, Hull JG, Kaufman PA, Li Z, Seville JL, Ahles TA, Kornblith AB, Hegel MT. Development and initial evaluation of a telephone-delivered, behavioral activation, and problem-solving treatment program to address functional goals of breast cancer survivors. J Psychosoc Oncol. 2015;33(2):199-218. doi: 10.1080/07347332.2014.1002659. Epub 2015 Feb 10. PMID 25668509